CLINICAL TRIAL: NCT05418465
Title: A Prospective, Open, Multicenter, Clinical Study of Huangqi Guizhi Wuwu Decoction in Treating Diabetic Nephropathy (Stage CKD2-4)
Brief Title: Huangqi Guizhi Wuwu Decoction in CKD Stage 2-4 Diabetic Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Principal Investigator, Ming Fang, Chief physician, The First Affiliated Hospital of Dalian Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PJ-KS-KY-2021-228(X2)
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Nephropathies
Keywords: Diabetic nephropathy,Huangqi Guizhi Wuwu Decoction (CKD2-4)
MeSH Terms: conditions — Diabetic Nephropathies | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huangqi Guizhi Wuwu decoction group (Experimental): Huangqi Guizhi Wuwu decoction
  Interventions: Drug: Huangqi Guizhi Wuwu decoction
- Dapagliflozin group (Active Comparator): Dapagliflozin
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Huangqi Guizhi Wuwu decoction — Huangqi Guizhi Wuwu decoction, 100ml at a time, 2 times a day. Oral administration.
  Arms: Huangqi Guizhi Wuwu decoction group
Drug: Dapagliflozin — Dapagliflozin, 10mg at a time, once a day. Oral administration.
  Arms: Dapagliflozin group

SUMMARY:
This is a prospective, open, multicenter clinical trial.The objective of this study is to evaluate the efficacy and safety of Huangqi Guizhi Wuwu Decoction in patients with CKD stage 2-4 diabetic nephropathy.

DETAILED DESCRIPTION:
The incidence rate of chronic kidney disease is 10.8% in China. The incidence rate of diabetic nephropathy has increased year by year, and now it has become the first cause of uremia. Therefore, the treatment of diabetic nephropathy can delay the progression of renal function and is of great value and significance in reducing uremia. Huangqi Guizhi Wuwu decoction is a traditional Chinese medicine decoction. Previous studies have shown that it is effective in the treatment of diabetic nephropathy. In this study, there were 2 hospitals participating in. We planned to enroll 100 participants, who will be divided into the Huangqi Guizhi Wuwu decoction group (experimental group) and the Dapagliflozin group (control group). All participants will take medication for 12 weeks, and investigators will follow up participates at weeks 0, 2,4, 6, 8,12.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as diabetic nephropathy
2. TCM syndrome differentiation is Qi deficiency and blood stasis type
3. Male or female, 18≤age≤75 4.25mL/（min.1.73m2）≤ eGFR<90mL/（min.1.73m2） 5.24-hour urine protein ration ≤3.5g/24h

6.The participants must be capable of understanding and comply with the protocol and sign a written informed consent document

Exclusion Criteria:

1. Exposure to immunosuppressors, glucocorticoid，without a one weeks washout period
2. Urinary tract infection (leukocytes in urinary sediment > 5 / HP)
3. Serum potassium > 5.5 mmol/L
4. Serum albumin < 30g/L
5. Pregnant or lactating women, and participants (including males) who were unable or unwilling to take adequate contraception during the study period
6. Having comorbidities that affect the progression of diabetic nephropathy (including but not limited to Malignant tumors, Systemic autoimmune diseases, Liver cirrhosis)
7. Participating in another clinical trial
8. Investigators do not think it suitable for a participant to join this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of change in Estimated Glomerular Filtration Rate (eGFR) compared to baseline | 12 weeks
  Events based on eGFR measure compared to baseline calculated using the CKD-EPI formula.

SECONDARY OUTCOMES:
Change in 24-hour urine protein ration from baseline. | Start of treatment until the end of the treatment for 12 weeks
  24-hour urinary protein quantification is being assessed once every 4 weeks for a total of 4 times during the whole study.

OTHER OUTCOMES:
Composite endpoint incidence | Start of treatment until the end of the treatment for 12 weeks
  The incidence of endpoint events：① eGFR decreased by 15% from baseline；② The incidence of doubling the quantitative change of 24-hour urinary protein (measured twice continuously).
Incidence of adverse reactions | Start of treatment until the end of the treatment for 12 weeks
  The proportion of patients with adverse reactions to the total population

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Dalian medical university, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided